CLINICAL TRIAL: NCT03398070
Title: Neuroimaging Biomarkers of Prognosis in Motor Functional Neurological Disorders
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David Lewis Perez, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 1K23MH111983-01A1 (NIH)
Record Dates: First submitted 2017-12-15; First posted 2018-01-12 (Actual); Results first posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Conversion Disorder
Keywords: Functional Neurological Disorder; Functional Movement Disorder; Psychogenic Nonepileptic Seizures; Functional Limb Weakness
MeSH Terms: conditions — Conversion Disorder; Psychogenic Nonepileptic Seizures | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Motor Functional Neurological Disorder.: The cohort will consist of patients with clinically established motor functional neurological disorder, which includes individuals with functional movement disorders, psychogenic nonepileptic seizures and functional limb weakness.
  Patients will be receiving the standard of care within the Massachusetts General Hospital (MGH) Functional Neurological Disorders Clinic.
  The updated standard of care that patient's receive in the MGH Functional Neurological Disorders Clinic includes the following:
  1. Delivery of a positive "rule-in" diagnosis of functional neurological disorder
  2. Individuals are provided with educational materials on functional neurological disorders
  3. Referred to physical therapy and/or occupational therapy as clinically indicated
  4. FND related cognitive behavioral therapy (CBT) referral when appropriate
  5. Psychotropic medication management based on standard psychiatric care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — The standard of care interventions for Functional Neurological Disorders (FND) include:
  1. delivery of a rule-in diagnosis
  2. providing educational materials
  3. referring to physical therapy (PT) and/or occupational therapy (OT) as clinically indicated
  4. referring to FND-related cognitive behavioral therapy (CBT)
  5. psychotropic medication management based on standard psychiatric care

SUMMARY:
Functional Neurological Disorder (FND/ Conversion Disorder) is a highly prevalent and disabling neuropsychiatric condition. Motor FND symptoms include Nonepileptic Seizures, Functional Movement Disorders and Functional Weakness. Clinical research across these motor FND subtypes, including research studies from the candidate's laboratory, suggest that these populations share many clinical and phenotypic similarities that warrant increased research integration. Furthermore, despite the prevalence of motor FND, little is known about the underlying pathophysiology of this condition, which is a prerequisite for the development of biologically informed prognostic and treatment response biomarkers. Across 3 published neurobiologically focused articles, the candidate proposed a framework through which to conceptualize motor FND. It is suggested that motor FND develops in the context of structural and functional alterations in neurocircuits mediating emotion awareness/expression, bodily awareness, viscerosomatic processing and behavioral regulation. The overall goal of this project is to comprehensively investigate structural and functional magnetic resonance imaging (MRI) biomarkers of prognosis across motor FND. Multimodal structural and functional MRI techniques (including voxel-based morphometry, cortical thickness, resting-state functional connectivity and diffusion tensor imaging tractography) will be used to systemically probe brain-prognosis relationships. Novel aspects of this proposal include the study of the full spectrum of motor FND, consistent with a trans-diagnostic approach.

DETAILED DESCRIPTION:
Functional Neurological Disorder (FND) (Conversion Disorder) is a poorly understood and prevalent somatoform disorder, making up 16% of outpatient neurology referrals. Patients with motor FND (mFND) are difficult to treat, result in major morbidity, and are costly to the US. An estimated $256 billion is spent annually treating this population. mFND includes Nonepileptic Seizures (NES), Functional Movement Disorders (FMD) and Functional Weakness (FW). An impediment to managing mFND is the lack of a neurobiological understanding for this disorder. The diagnosis of mFND is currently based on qualitative aspects of behaviors, which may be difficult to interpret, and the absence of findings characteristic of other neuropsychiatric disorders on laboratory studies such as electroencephalography (EEG) and magnetic resonance imaging (MRI).

A major step forward would be the identification of neuroimaging biomarkers for mFND. mFND is understudied compared to other disorders, but recent studies point to distributed neurocircuit alterations associated with mFND. This project aims to advance our biological understanding of mFND by investigating neuroimaging biomarkers linked to prognosis. An improved understanding of the pathophysiology of mFND will provide a critical step in elucidating diagnostic, prognostic and treatment response biomarkers.

Aim:

Identify structural and functional biomarkers of prognosis at 6-months in patients with motor functional neurological disorders receiving an updated standard of care.

H1: Favorable mFND prognosis at 6 months post initial evaluation will be predicted by the degree of preserved baseline gray matter in limbic-paralimbic regions, particularly those part of the salience network.

H2: Favorable mFND prognosis at 6 months post initial evaluation will be predicted by the degree of preserved baseline resting-state functional connectivity in limbic/paralimbic areas, particularly those part of the salience network.

H3: Favorable mFND prognosis at 6 months will correlate with the degree of preserved baseline cingulum bundle and cingulum-insular tract integrity.

ELIGIBILITY:
Inclusion Criteria:

* clinically established motor functional neurological disorder, including individuals with functional movement disorders, functional limb weakness and psychogenic nonepileptic seizures

Exclusion Criteria:

* active suicidality
* major medical/neurological comorbidities with known central nervous system (CNS) consequences
* active drug use or alcohol dependence
* known history of a primary psychotic disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment will occur from patients receiving care in the Massachusetts General Hospital (MGH) Functional Neurological Disorders Clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Diez I, Ortiz-Teran L, Williams B, Jalilianhasanpour R, Ospina JP, Dickerson BC, Keshavan MS, LaFrance WC Jr, Sepulcre J, Perez DL. Corticolimbic fast-tracking: enhanced multimodal integration in functional neurological disorder. J Neurol Neurosurg Psychiatry. 2019 Aug;90(8):929-938. doi: 10.1136/jnnp-2018-319657. Epub 2019 Mar 8. PMID 30850473
- [Result] Perez DL, Williams B, Matin N, Mello J, Dickerson BC, LaFrance WC Jr, Keshavan MS. Anterior hippocampal grey matter predicts mental health outcome in functional neurological disorders: an exploratory pilot study. J Neurol Neurosurg Psychiatry. 2018 Nov;89(11):1221-1224. doi: 10.1136/jnnp-2017-317305. Epub 2018 Jan 11. No abstract available. PMID 29326291
- See also: See Figure 5 for relevant results — https://jnnp.bmj.com/content/90/8/929.long
- See also: See Figure 1 for relevant results — https://jnnp.bmj.com/content/89/11/1221.long

RESULTS

PARTICIPANT FLOW:
Groups:
- Motor Functional Neurological Disorder.: The cohort will consist of patients with clinically established motor functional neurological disorder, which includes individuals with functional movement disorders, psychogenic nonepileptic seizures and functional limb weakness.
  Patients will be receiving the standard of care within the Massachusetts General Hospital (MGH) Functional Neurological Disorders Clinic.
  The updated standard of care that patient's receive in the MGH Functional Neurological Disorders Clinic includes the following:
  1. Delivery of a positive "rule-in" diagnosis of functional neurological disorder
  2. Individuals are provided with educational materials on functional neurological disorders
  3. Referred to physical therapy and/or occupational therapy as clinically indicated
  4. FND related cognitive behavioral therapy (CBT) referral when appropriate
  5. Psychotropic medication management based on standard psychiatric care
  Standard of Care: The standard of care interventions for Functional Neurological Disorders (FND) include:
  1. delivery of a rule-in diagnosis
  2. providing educational materials
  3. referring to physical therapy (PT) and/or occupational therapy (OT) as clinically indicated
  4. referring to FND-related cognitive behavioral therapy (CBT)
  5. psychotropic medication management based on standard psychiatric care
Period: Overall Study
Arm/Group | Motor Functional Neurological Disorder.
Started | 30
Completed | 22
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Motor Functional Neurological Disorder.
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Gray Matter Volume Biomarkers of 6 Month Prognosis as Measured by Voxel Based Morphometry - Within Group Comparison
Description: Correcting for multiple comparisons in structural analyses, baseline structural grey matter volumes in limbic/paralimbic regions (particularly those affiliated with the salience network), would relate to clinical outcome in individuals receiving the standard of care at 6 months. Analyses reported refer to change in either mental health or physical health scores and baseline gray matter volume. The number presented is the peak voxel z-score as also reported in Supplementary Table 4 of the published manuscript.
  Z-scores are presented in absolute values (with the lowest value being 0). A higher z-score represents a stronger correlation between a given gray matter volume value (at the peak voxel) and the measure of interest (in case mental health or physical health scores). The entry under "row title" specifies if the association is a "positive" vs a "negative" association.
Time Frame: baseline and 6 months
Population: For this study, of an initially enrolled 30 participants, 22 provided followup data.
Measure: Number; unit: peak voxel z-score
Arm/Group | Motor Functional Neurological Disorder.
Number analyzed (Participants) | 22
peak voxel z-score
  ∆SF-36 Mental Health Positive Associations: R supplementary motor area (6): 10mm, -16mm, 75mm | 4.18
  ∆SF-36 Mental Health Positive Associations: R superior frontal gyrus (6): 18mm, -7mm, 72mm | 3.27
  ∆SF-36 Mental Health Positive Associations: R middle cingulate gyrus (24): 3mm, 12mm, 43mm | 3.85
  ∆SF-36 Mental Health Positive Associations: L anterior hippocampus: -34mm, -16mm, -15mm | 3.76
  ∆SF-36 Mental Health Positive Associations: L middle frontal gyrus (46): -33mm, 26mm, 40mm | 3.61
  ∆SF-36 Physical Health Positive Associations: R frontopolar cortex (10): 10mm, 62mm, 4mm | 3.90
  ∆SF-36 Physical Health Negative Associations: R superior/middle frontal gyrus (9): 22mm, 24mm, 37mm | 4.40
  ∆SF-36 Physical Health Negative Associations: L superior occipital gyrus (19): -10mm, -82mm, 45mm | 3.80
  ∆SF-36 Physical Health Negative Associations: L superior occipital gyrus (19): -18mm, -78mm, 42mm | 3.70

2. Primary Outcome: Resting State Functional Connectivity Strength Biomarkers of 6 Month Prognosis - Within Group Comparison
Description: Correcting for multiple comparisons in resting state connectivity analyses, baseline functional connectivity strength (t-statistic scores) across limbic/paralimbic regions (particularly those affiliated with the salience network), would relate to clinical outcome in individuals receiving the standard of care at 6 months. Here, we tested if link-step connectivity from primary motor areas or amygdala nuclei related to change in clinical outcome. Specifically, we are providing the t-statistic for the connectivity strength between left centromedial amygdala to right anterior insula.
  Functional connectivity strength is based on the correlation of low frequency brain oscillations measured at rest. A large t-statistic value reflects greater connectivity between brain voxels.
Time Frame: baseline and 6 months
Population: For this study, of an initially enrolled 30 participants, 22 provided followup data.
Measure: Number; unit: t-statistic
Arm/Group | Motor Functional Neurological Disorder.
Number analyzed (Participants) | 22
t-statistic | 4.58

3. Primary Outcome: The Integrity of Specific White Matter Tracts (Fractional Anisotropy) as Measured by Diffusion Tensor Imaging (DTI) Tractography Will Relate to 6-month Prognosis
Description: Baseline integrity of the cingulum bundle and cingulate-insular tracts, as measured by fractional anisotropy, would relate to 6 month prognosis in patients with Functional Neurological Disorders (FND) receiving the standard of care.
  Outcome was not assessed - no time to analyze data given prior challenges with the pandemic. Unable to report data in any table as the white matter images have not been analyzed.
Time Frame: baseline and 6 months
Population: we focused on our T1-weighted structural and functional connectivity analyses during this K23 grant period.
Arm/Group | Motor Functional Neurological Disorder.
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 5 years of research funding
Arm/Group | Motor Functional Neurological Disorder.
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

LIMITATIONS AND CAVEATS:
Limitations include a modest sample size, patient heterogeneity, medication use, reliance on self-report measures and that management was not restricted to one institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT03398070/Prot_SAP_001.pdf